CLINICAL TRIAL: NCT01632046
Title: Randomized, Long-Term Administration of pH-Neutral PD Solutions Containing Lactate (BALANCE) or Bicarbonate (BICAVERA) in Children
Brief Title: Administration of pH-Neutral Peritoneal Dialysis Solutions Containing Lactate or Bicarbonate in Children
Acronym: BIOKID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Claus Peter Schmitt, M.D., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOKID 04 EU; University of Heidelberg (Other: Investigator Initiated Trial, University of Heidelberg)
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Renal Failure; Peritoneal Membrane Disorder
Keywords: peritoneal dialysis; bicarbonate/lactate buffer; peritoneal transport capacity; ultrafiltration; children
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BicaVera, dialysis (Active Comparator): Two Parallel arms. If patient randomised to the BicaVera arm he will be dialysed with bicarbonate based PD fluid (BicaVera) for 10 months. Dialysis prescription is determined according to clinical needs, dialysate glucose concentrations are 1.5, 2.3 and 4.25 %.
  Interventions: Drug: lactate and bicarbonate buffered dialysis solutions
- Balance, dialysis (Active Comparator): If patient is randomised to the Balance arm, he will be dialysed with lactate based PD fluid (Balance) for 10 months. Dialysis prescription is determined according to clinical needs, dialysate glucose concentrations are 1.5, 2.3 and 4.25 %.
  Interventions: Drug: lactate and bicarbonate buffered dialysis solutions

INTERVENTIONS:
Drug: lactate and bicarbonate buffered dialysis solutions — Either PD-solution will be applied. Number of cycles and glucose concentration will be varied according to clinical needs. Sleep Safe system will be used and connected to Sleep Safe Cyclers in patient on CCPD.
  Other Names: BicaVera; Balance

SUMMARY:
Peritoneal Dialysis (PD) is the preferred treatment modality in children with end-stage renal disease. Unfortunately progressive alterations of the peritoneal membrane occur with time on PD, leading to a continuous loss of peritoneal transport function. Recently, double-chambered PD solutions with less Glucose Degradation Products (GDPs) and neutral pH have been approved for the European market. Short term administration suggests comparable clearance rates compared with conventional solutions. In vitro studies demonstrate an improved local immune defense system. To compensate for metabolic acidosis, the available solutions either contain lactate or bicarbonate, the impact of either buffer on long term acidosis control and peritoneal membrane integrity, however, is unknown.

The prospective, European multi-center study will provide the first long term administration of pH neutral, low GDP solutions in children. 60 children will randomly be treated with a bicarbonate (BicaVera) and a lactate based solution (Balance), respectively. The primary end point will be the effect of either PD-solution on peritoneal transport characteristics (D/P Creatinine). Secondary end-points will be the effects on ultrafiltration capacity, acid-base balance, peritoneal morphology, incidence and severity of peritonitis, and on surrogate parameters of biocompatibility and carbonyl stress. Moreover, potential genetic determinants of the peritoneal transporter status and of the continued morphological transformation of the peritoneum will be assessed.

After a 2 month run-in period, using a conventional, acidic, single-chambered PD-solution, the patients will be randomized to a 10 month study period using BicaVera and Balance, respectively. Dialysis regime and follow up in the out-patient clinic will be performed according to clinical needs (every 4 weeks); episodes of peritonitis will be treated according to international guidelines. Bicarbonate supplements will be prescribed at a dose of 0.5 mmol/kg *d, if blood bicarbonate levels fall below 17 mmol/l. PD adequacy will be verified by routine, monthly venous blood sampling and a capillary blood gas analysis. 2-5 ml of blood will be drawn for analysis of relevant gene polymorphisms. At study entry, after 3, 6 and 10 months, a 24h dialysate- and urine collection, a peritoneal equilibration test an intraperitoneal pressure measurement will be performed. Peritoneal biopsies will be obtained at any time of abdominal surgery. Adverse events will be screened meticulously. The trial will be carried out in accordance with the German medicines act (AMG) and other local requirements, with particular reference to the ICH guidelines for Good Clinical Practice, and the declaration of Helsinki. At study end, the patients will decide together with the responsible physician which PD-fluid should be used further one.

DETAILED DESCRIPTION:
For details please see Nau B, Schmitt CP et al; BMC Nephrol. 2004 Oct 14;5:14.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 1 months to 21 years of age (newborns excluded)
* CAPD or CCPD for end stage renal disease
* Dwell volume ~ 1100ml/m² body surface area
* Last peritonitis at least 3 weeks ago
* Written informed consent

Exclusion Criteria:

* Reduced efficiency of peritoneal dialysis due to anatomic anomalies or intraperitoneal adhesions
* Uncontrolled hyperphosphatemia
* Participation in a clinical trial with an investigational drug within one month prior start of study. Prior participation in this trial
* Suspicion of drug abuse
* Severe pulmonary, cardiac or hepatic disease/insufficiency
* Any kind of malignancy

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of a lactate based and a bicarbonate based double-chambered, pH-neutral PD solution on peritoneal transport capacity in children. | 2 months run in 10 months study period
  Following a two months run in period patients are randomized to either lactate or bicarbonate buffered PD solution. The primary outcome measure is dialysate over plasma creatinine as a measure of peritoneral transport efficacy. It will be determined at 0, 3, 6 and 10 months.

SECONDARY OUTCOMES:
Ultrafiltration | 2 months run in 10 months observation
  The ultrafiltration is recorded daily by the caretakers, mean weakly ultrafiltration will be analysed. (Further outcome measures include the effect of either PD solution on acid-base balance, incidence and severity of peritonitis, and on surrogate parameters of biocompatibility and carbonyl stress).

CONTACTS AND LOCATIONS:
Overall Officials: Claus P Schmitt, M.D., Principal Investigator — University of Heidelberg, Center for Pediatric and Adolescent Medicine
Locations (7):
- University Children's Hospital, Vienna, Austria
- University Children's Hospital, Helsinki, Finland
- University Children's Hospital, Strasbourg, France
- Germany (3):
  - University Children's Hospital, Essen
  - University Children´s Hospital, Hamburg
  - University Children's Hospital, Jena
- University Children's Hospital, Milan, Italy

REFERENCES:
- [Background] Nau B, Schmitt CP, Almeida M, Arbeiter K, Ardissino G, Bonzel KE, Edefonti A, Fischbach M, Haluany K, Misselwitz J, Kemper MJ, Ronnholm K, Wygoda S, Schaefer F; European Pediatric Peritoneal Dialysis Study Group. BIOKID: randomized controlled trial comparing bicarbonate and lactate buffer in biocompatible peritoneal dialysis solutions in children [ISRCTN81137991]. BMC Nephrol. 2004 Oct 14;5:14. doi: 10.1186/1471-2369-5-14. PMID 15485574
- [Derived] Schmitt CP, Nau B, Gemulla G, Bonzel KE, Holtta T, Testa S, Fischbach M, John U, Kemper MJ, Sander A, Arbeiter K, Schaefer F. Effect of the dialysis fluid buffer on peritoneal membrane function in children. Clin J Am Soc Nephrol. 2013 Jan;8(1):108-15. doi: 10.2215/CJN.00690112. Epub 2012 Nov 2. PMID 23124784